CLINICAL TRIAL: NCT06957379
Title: A Phase II Clinical Trial of the Safety and Efficacy of Sirolimus for Injection (Albumin-bound) in Combination With Endocrine Therapy for the Treatment of HR-positive, HER2-negative Patients With Advanced Breast Cancer Who Have Failed Standard Therapy
Brief Title: Sirolimus for Injection (Albumin-bound) in Combination With Endocrine Therapy for HR+/HER2- Advanced/Metastatic Breast Cancer Patients Who Have Failed Standard Therapy
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HB1901-005
Record Dates: First submitted 2025-04-26; First posted 2025-05-04 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: HR+/HER2- Advanced/Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Letrozole; Anastrozole; exemestane; Fulvestrant; Sirolimus; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sirolimus for Injection (Albumin-bound) Combined with Fulvestrant or Aromatase Inhibitor (Experimental): A: Sirolimus for Injection (Albumin-bound) Combined with Fulvestrant; B: Sirolimus for Injection (Albumin-bound) Combined with Exemestane，or Letrozole，or Anastrozole.
  Interventions: Drug: Letrozole; Drug: Anastrozole; Drug: Exemestane; Drug: Fulvestrant; Drug: Sirolimus for Injection (Albumin-bound)

INTERVENTIONS:
Drug: Letrozole — Oral administration at a dose of 2.5 mg once daily for a 4-week cycle
Drug: Anastrozole — Oral administration at a dose of 1 mg once daily for a 4-week cycle
Drug: Exemestane — Oral administration at a dose of 25 mg once daily with a meal every 4 weeks
Drug: Fulvestrant — Fulvestrant: IM injection, 500 mg, on day 1 and day 15 of Cycle 1, and then on day 1 of each cycle thereafter, 4 weeks per treatment cycle
Drug: Sirolimus for Injection (Albumin-bound) — IV infusion, every 2 weeks, 4 weeks per treatment cycle

SUMMARY:
This study is a multicenter, open, non-randomized phase II clinical trial consisting of a safety introduction phase followed by a single-arm phase 2 phase. This phase II trial enrolled patients with HR+/HER2- advanced breast cancer who had failed aromatase inhibitor (AI)/fulvestrant ± CDK4/6i. Pts failing prior AI ± CDK4/6i received nab-Sirolimus + fulvestrant, while those failing fulvestrant ± CDK4/6i received nab-Sirolimus + AI.

ELIGIBILITY:
Inclusion Criteria:

* 1. Aged 18 or above, regardless of gender; female patients must be postmenopausal, or premenopausal/perimenopausal.
* 2. Pathologically confirmed HR+, HER2- breast cancer.
* 3. Patients who have failed prior treatment with AI or fulvestrant with or without CDK4/6 inhibitors.
* 4. No more than 3 lines of chemotherapy for inoperable locally advanced or metastatic disease.
* 5. At least one measurable lesion according to RECIST 1.1 criteria. Patients with bone lesions only may be eligible.
* 6. ECOG performance status score of 0-1.
* 7. Investigator-assessed life expectancy ≥3 months.
* 8. Adequate organ and bone marrow function.
* 9. Baseline fasting serum triglyceride <300mg/dL or 3.42mmol/L, fasting serum cholesterol <350mg/dL or 9.07mmol/L
* 10. The baseline fasting plasma glucose (FPG) ˂ 7.8 mmol/L and glycosylated hemoglobin (HbA1c) ˂ 8%
* 11. Premenopausal female patients using LHRH agonists to suppress ovarian function must agree to use two acceptable forms of highly effective contraception during the study and for 6 months after stopping study treatment; female patients of childbearing potential must have a negative pregnancy test before starting study treatment and must not be breastfeeding.
* 12. Male patients must agree to use barrier contraception (i.e., condoms) during the study and for 6 months after stopping study treatment; for men with future fertility plans, sperm freezing is recommended before starting study treatment.
* 13. Participants must provide informed consent before the trial and voluntarily sign the written ICF.

Exclusion Criteria:

* 1. Previous pathological diagnosis of HER2-positive breast cancer.
* 2. Patients judged by the investigator to be unsuitable for endocrine therapy.
* 3. Patients who have previously received PI3K/AKT/mTOR inhibitors.
* 4. Received chemotherapy, radiotherapy, biological therapy, targeted therapy, immunotherapy, or other anti-tumor treatments within 4 weeks before randomization.
* 5. Received other unapproved investigational drugs within 4 weeks before randomization.
* 6. Underwent major surgery within 4 weeks before randomization or has not fully recovered from any previous invasive procedures.
* 7. Received systemic glucocorticoids (prednisone >10 mg/day or equivalent) or other immunosuppressive treatments within 2 weeks before randomization.
* 8. Had an infection within 2 weeks before randomization requiring systemic (oral or IV) anti-infective treatment (uncomplicated urinary tract infections or upper respiratory tract infections excluded).
* 9. Received inactivated or live attenuated vaccines or COVID-19 vaccines within 4 weeks before randomization.
* 10. Used strong inhibitors or inducers of CYP3A4 hepatic metabolic enzymes within 2 weeks before randomization or still need to continue using such drugs.
* 11. Diagnosed with other malignancies within 5 years before randomization.
* 12. Suffering from severe cardiovascular or cerebrovascular diseases.
* 13. Adverse reactions from previous anti-tumor treatments have not recovered to CTCAE 5.0 grade ≤1.
* 14. Active leptomeningeal disease or poorly controlled central nervous system metastases.
* 15. Presence of pleural/abdominal effusion or pericardial effusion with clinical symptoms or requiring symptomatic treatment.
* 16. Known bleeding tendency (constitution) or coagulation disorders.
* 17. History of severe lung diseases such as interstitial lung disease and/or pneumonia, pulmonary hypertension, or radiation pneumonitis requiring glucocorticoid treatment.
* 18. Known hypersensitivity or intolerance to any component of the study drug or its excipients, or LHRH agonists (if applicable).
* 19. History of autoimmune diseases (except tuberous sclerosis), immunodeficiency diseases, including HIV-positive, or other acquired or congenital immunodeficiency diseases, or organ transplant history.
* 20. Active HBV, HCV, syphilis, or tuberculosis infection.
* 21. Other conditions judged by the investigator to be unsuitable for participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2024-02-29 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Up to ~24 months

SECONDARY OUTCOMES:
Disease Control Rate (DCR） | Up to ~36 months
Duration of Response (DoR) | Up to ~24 months
Progression-Free Survival (PFS) | Up to ~24 months
Overall Survivial (OS) | Up to ~24 months
Safety and Tolerability :the incidence and severity of Treatment Emergent Adverse Events（TEAEs）and Treatment-Related Adverse Events（TRAEs） | Up to ~24 months
PK parameter: the concentration of sirolimus | Up to ~24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China